CLINICAL TRIAL: NCT05794438
Title: Gamified Adaptive Approach Bias Modification on Individuals With Methamphetamine Use History
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS001
Record Dates: First submitted 2023-03-06; First posted 2023-04-03 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Addiction, Substance
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive Approach Bias Modification (Experimental)
  Interventions: Behavioral: Adaptive Approach Bias Modification
- Static Approach Bias Modification (Experimental)
  Interventions: Behavioral: Static Approach Bias Modification
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Static Approach Bias Modification — In the static approach bias modification, users were instructed to swipe upward when they see portrait format images and swipe downward when they see landscape format images. A shrinking animation comes after swiping upward to simulate the visual effect of moving away (approach), and a growing animation comes after swiping downward to simulate the visual effect of moving towards (avoidance). Two types of images, namely drug-related and non-drug-related, were used in the training. The drug-related images were related to methamphetamine (methamphetamine crystals, powders, and paraphernalia), and the non-drug-related images were related to healthy lifestyles (wealth, sports, gourmet, family activities, etc).
  Arms: Static Approach Bias Modification
Behavioral: Adaptive Approach Bias Modification — In the adaptive approach bias modification, users were instructed to swipe upward when they see portrait format images and swipe downward when they see landscape format images. A shrinking animation comes after swiping upward to simulate the visual effect of moving away (approach), and a growing animation comes after swiping downward to simulate the visual effect of moving towards (avoidance). Two types of images, namely drug-related and non-drug-related, were used in the training. The drug-related images were related to methamphetamine (methamphetamine crystals, powders, and paraphernalia), and the non-drug-related images were related to healthy lifestyles (wealth, sports, gourmet, family activities, etc). An algorithm continuously monitors the performance of the user and adjusts the ratio of congruent and incongruent trials accordingly to attain a desired difficulty curve.
  Arms: Adaptive Approach Bias Modification

SUMMARY:
A randomized controlled trial will be conducted to investigate whether a proposed algorithm that adjusts the congruency ratio based on the user's performance and difficulty can enhance the effectiveness of approach bias modification. Methamphetamine users will be recruited and randomized into an algorithm group, a standard group, and a control group.

DETAILED DESCRIPTION:
To assess the efficacy of an adaptive approach bias modification (A-ApBM) paradigm with gamified designs and dynamic difficulty adjustments in reducing cue-induced craving in individuals with methamphetamine use history. DESIGN: Randomized controlled trial with three study groups: Adaptive ApBM (A-ApBM), Static ApBM (S-ApBM), and control. A-ApBM and S-ApBM groups engaged in ApBM training using a smartphone application for four weeks. A-ApBM used an adaptive algorithm to dynamically adjust the difficulty level based on individual performance, while S-ApBM had a static difficulty level. Cue-induced craving scores were assessed using a visual analog scale at baseline, post-intervention, and at week-16 follow-up.

ELIGIBILITY:
Inclusion Criteria:

• having a history of methamphetamine use of at least one year

Exclusion Criteria:

* could not fluently operate an Android or an iOS smartphone
* having mental health conditions other than MUD

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Cue induced craving for methamphetamine | Baseline
  The cue-induced craving was assessed by showing the participants images related to methamphetamine (methamphetamine crystals, powders, and paraphernalia) on a smartphone and asking them to rate their cravings on a 0-10 visual analog scale (0 being least craved and 10 being most craved).
Cue induced craving for methamphetamine | Immediately Post-intervention
  The cue-induced craving was assessed by showing the participants images related to methamphetamine (methamphetamine crystals, powders, and paraphernalia) on a smartphone and asking them to rate their cravings on a 0-10 visual analog scale (0 being least craved and 10 being most craved).
Cue induced craving for methamphetamine | 16 week from baseline assesment
  The cue-induced craving was assessed by showing the participants images related to methamphetamine (methamphetamine crystals, powders, and paraphernalia) on a smartphone and asking them to rate their cravings on a 0-10 visual analog scale (0 being least craved and 10 being most craved).

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Gao Ping Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Han Zhou Street Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Jin Lun Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Jin Yan Street Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Jin Yu Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Lian Shan Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Nan Feng Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - San Shui Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Sanxingdui Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - SixTwentySix Service Center, Luo Cheng Street, Guanghan City, Luocheng, Sichuan
  - Xiang Yang Town Community Drug Rehabilitation Center, Luocheng, Sichuan
  - Xiao Han Town Community Drug Rehabilitation Center, Luocheng, Sichuan